CLINICAL TRIAL: NCT06024005
Title: A Prospective Randomized Controlled Trial: Comparison of the Transcutaneous Posterior Tibial Nerve Stimulation and Oral Solifenacin Treatments' Effects in Women Between 18-80 Years Old Who Have Overactive Bladder
Brief Title: Comparison of the Transcutaneous Tibial Nerve Stimulation and Drug Treatment' Effects in Women With Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ahmet Ozgur Yeniel, Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTNS for OAB
Record Dates: First submitted 2023-07-02; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome
Keywords: Overactive Bladder; Transcutaneous Electric Nerve Stimulation; Neuromodulation; Urge Urinary Incontinence; Quality of Life
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Group (Active Comparator): Transcutaneous device group with Urostim 2
  Interventions: Device: Transcutaneous Posterior Tibial Nerve Stimulation (TTNS)
- Drug Group (Active Comparator): Drug Group with Kinzy 5 mg
  Interventions: Drug: Oral Solifenacin 5mg

INTERVENTIONS:
Drug: Oral Solifenacin 5mg — Oral solifenacin (Kinzy 5mg) use once a day for 6 weeks
  Other Names: Kinzy 5mg
  Arms: Drug Group
Device: Transcutaneous Posterior Tibial Nerve Stimulation (TTNS) — Application of TTNS twice a week for 6 weeks, with each session for 30 minutes
  Other Names: Urostim 2
  Arms: Device Group

SUMMARY:
Overactive bladder (OAB) syndrome is a symptom complex characterized by sudden urgency, frequent urination, nocturia, and urge incontinence without any identifiable organic cause, significantly impacting the quality of life. One of the most prominent symptoms is the urgency to urinate accompanied by a sudden sensation of bladder fullness.

There are various treatment options available for managing OAB, including conservative therapy, pharmacotherapy, and surgical management. High-level evidence supports solifenacin as the standard medical treatment for OAB, offering advantages such as not being affected by food intake, efficacy regardless of gender, and high bioavailability. However, it is known to cause discontinuation of treatment in many cases due to the occurrence of side effects. Posterior tibial nerve stimulation (PTNS) is a neuromodulation technique that has been internationally recognized and proven effective in the treatment of OAB, providing several advantages. It can be applied through two methods: percutaneous (PTNS) and transcutaneous (TTNS). PTNS is an invasive method that requires specialized equipment and a trained healthcare professional, which limits its routine use due to treatment costs.

In the literature, it is stated that in the treatment of OAB, alone or combined PTNS applications are superior to drug monotherapies, but there are limited studies on this subject. Therefore, the study aim was to compare the efficacy, side effects and quality of life of solifenacin and TTNS.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 34 female patients with OAB were enrolled in the study. The patients were randomly divided into two groups, with 17 individuals in each group. Patients with odd case numbers were assigned to the Oral Solifenacin group, while those with even case numbers were assigned to the TTNS group.

Prior to treatment, the sociodemographic characteristics, birth history, and past treatment information of all participants were recorded. Basic urogynecological evaluation, pelvic floor ultrasound, and urine culture were performed. To assess symptoms and quality of life, the Overactive Bladder Assessment Form (OAB-V8), Incontinence Quality of Life Scale (I-QQL), Incontinence Impact Questionnaire (IIQ-7), Urogenital Distress Inventory (UDI-6), and a three-day bladder diary were used. After 6 weeks of treatment, all evaluations were repeated. The treatment regimen consisted of once-daily oral solifenacin for the medication group and 2 sessions per week, 30 minutes per session, for 12 sessions using the Urostim-2 device for the TTNS group. The stimulation intensity was increased until a motor or sensory response was obtained, and the threshold value was determined. The entire TTNS procedure was performed under the supervision of an expert physician at the Urogynecology Outpatient Clinic of Ege University Hospital. Statistical analysis was conducted using SPSS 20.0.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with a diagnosis of OAB and unresponsive to first-line treatment,
* Absence of genito-urinary system malformations that may cause pollacullaire,
* Volunteering to participate in the research,
* To be literate in Turkish

Exclusion Criteria:

* Having a urinary tract infection,
* Having pelvic organ prolapse greater than stage 2,
* To be diagnosed with stress type urinary incontinence,
* Having narrow-angle glaucoma, myasthenia gravis and severe gastro-intestinal diseases,
* Patients undergoing hemodialysis,
* Having severe liver or kidney failure,
* Pregnancy,
* Having a pacemaker
* Presence of epilepsy,
* The presence of built-in metal in the ankle
* Open ankle wound

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Number of Total Daily Incontinence Episodes | 6 weeks
  It was obtained using a three-day bladder diary. Objective. Meaningful for patients. Correlates with patients' daily activities. It may not be directly related to the severity of urine leakage. Subject to variability. Requires patient compliance. Day and night urine leakages were recorded separately by the patient for three days. The mean total score for a day was calculated.
Evaluation of Quality of Life | 6 weeks
  The Incontinence Quality of Life Scale (I-QOL), consisting of 22 questions, was used to analyze the improvement in quality of life. It is a validated questionnaire. Higher scores indicate a better level of quality of life compared to lower scores. It is meaningful for patients. It is standardized. It takes into account the patient's daily activities. Subjective. Subject to variability. Not correlated with the severity of urine leakage.

SECONDARY OUTCOMES:
Symptom Assessment | 6 weeks
  Overactive Bladder Assessment Form (OAB-V8), was used for symptomatic evaluation and to assess the impact of symptoms on quality of life. It is a validated questionnaire. A higher score means a worse outcome. Meaningful for patients. It is standardized. The patient's daily activities are taken into account. Subjective. Subject to variability. Not correlated with the severity of urine leakage.
Symptom Assessment | 6 weeks
  Urogenital Distress Inventory (UDI-6), was used for symptomatic evaluation and to assess the impact of symptoms on quality of life. It is a validated questionnaire. A lesser score means a better outcome. Meaningful for patients. It is standardized. The patient's daily activities are taken into account. Subjective. Subject to variability. Not correlated with the severity of urine leakage.
Symptom Assessment | 6 weeks
  Incontinence Impact Questionnaire (IIQ-7), was used for symptomatic evaluation and to assess the impact of symptoms on quality of life. It is a validated questionnaire. A lesser score means a better outcome. Meaningful for patients. It is standardized. The patient's daily activities are taken into account. Subjective. Subject to variability. Not correlated with the severity of urine leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Ozgur OY Yeniel, Principal Investigator — Ege University School of Medicine, Department of Obstetrics and Gynecology,
Locations (1):
- Ege University, School of Medicine, Department of Obstetrics and Gynecology, Izmir, Turkey (Türkiye)